CLINICAL TRIAL: NCT03110614
Title: Diastolic Dysfunction and Pauci-inflammatory Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Diastolic Dysfunction and Pauci-inflammatory Acute Exacerbations of COPD
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Surya P Bhatt, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F121120003; K23HL133438-01 (NIH)
Record Dates: First submitted 2017-03-15; First posted 2017-04-12 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Diastolic Dysfunction
Keywords: COPD; acute; exacerbation; lung ultrasound
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Exhaled breath condensate for inflammatory markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective study to determine the relationships between pauci-inflammatory exacerbations and diastolic dysfunction, and their implications in hospitalized patients with acute exacerbations of COPD. To assess changes within subjects from stable to acute phase, a number of comparisons will be made in subjects enrolled during acute exacerbation with similar measurements made in the stable phase after recovery from exacerbation after at least 35 days from index hospitalization or prior exacerbation.

DETAILED DESCRIPTION:
Informed consent will be obtained within the first 24 hours of admission. Written informed consent will be obtained from the subject or a legally authorized representative.

Visit Schedule:

V1 (Day 0 of Hospitalization):

Demographic and clinical information including age, gender, race, smoking status, number of pack-years of smoking, body mass index, waist hip circumference, co-morbidities such as diabetes mellitus, hypertension, hyperlipidemia, depression, coronary artery disease and chronic kidney disease, history of previous exacerbations, detailed occupation history, and detailed medication history with emphasis on cardiovascular medications will be conducted. The COPD Assessment Test (CAT) questionnaire and the modified Medical Research Council (mMRC) assessment will be administered. Bed-side spirometry will be conducted. Blood will be drawn for lab tests (about 30 mL or 6 teaspoons). Electrocardiography (ECG), lung ultrasound and echocardiography will be performed.

V2 (hospital discharge day or day 3 of hospitalization whichever is earlier):

Blood will be drawn for lab test- CRP only ( about 5mL or 1 teaspoon). Participant will be scheduled for a follow-up visit at the Lung Health Center.

V3 (Day 35- Follow-up visit at Lung Health Center):

The COPD Assessment Test (CAT) questionnaire and the modified Medical Research Council (mMRC) assessment will be administered. The following Pulmonary Function Tests will be conducted: Spirometry, lung Volumes and DLCO. Six-minute walk test will be conducted. Blood will be drawn for lab tests (about 30 mL or 6 teaspoons). Electrocardiography, lung ultrasound and echocardiography will be performed.

Telephone follow-up: The participant will be called once every 6 months for one year, to ask about COPD symptoms.

Description of procedures:

Questionnaires:

Dyspnea: will be assessed using the modified Medical Research Council (mMRC). The mMRC scale is a simple grading system to assess a patient's level of dyspnea, ranging from 0 for minimal to 4 for severe dyspnea.

COPD related Quality of life: will be assessed using the COPD Assessment Test (CAT) The CAT questionnaire consists of 8 simple questions which are graded from 0 to 5. The total score can range from 0 to 40. A change of 2 units is considered clinically significant (minimal clinically important difference).

Pulmonary Function Tests (PFTs):

Bedside spirometry will be performed using a handheld spirometer, and the following parameters will be recorded: forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), FEV1/FVC ratio , forced expiratory flow in the middle 25 to 75% of flow (FEF25-75%), inspiratory capacity (IC), and peak expiratory flow rate (PEFR). A subsequent full set of pulmonary function tests will be obtained in the recovery phase on day 35 using a hand held spirometer and body plethysmography. This will include FEV1 , FVC, FEV1/FVC, FEF25-75%, IC, PEFR, total lung capacity (TLC), residual volume (RV), and diffusing capacity of carbon monoxide (DLCO).

Blood: will be collected to measure markers of systemic inflammation such as C-reactive protein (CRP), fibrinogen, IL-6 and TNF-alpha, and measures of cardiac function such as troponin and brain natriuretic peptide (BNP).

Six-Minute Walk Test: The 6 minute walk test measures the mean distance walked on a 100 meter straight, hard-surfaced coarse in 6 minutes while being continuously monitored by the study coordinator.

Ultrasound of lungs: B mode ultrasonography will be used to assess pulmonary congestion.

Echocardiography: Parameters of systolic and diastolic function will be assessed using 2D and Doppler echocardiography using standard echo windows.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older
* Patients admitted to the general medicine or pulmonary floors, or the medical intensive care unit with a primary diagnosis of acute exacerbation of COPD will be eligible for the study.

Exclusion Criteria:

* Patients with a secondary diagnosis of congestive heart failure and other respiratory conditions that the investigator's deem could confound the diagnosis including but not limited to pneumonia, bronchiectasis and lung cancer will be excluded.
* Pregnant or breastfeeding women will be excluded.
* Patients with conditions that preclude an adequate echocardiogram such as hemodynamically significant arrhythmias will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with acute exacerbations of COPD will be approached for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Difference in the proportion of diastolic dysfunction in pauci-inflammatory exacerbations vs. inflammatory exacerbations | at baseline (at time of hospitalization)
  We will estimate the frequency of diastolic dysfunction on echocardiogram in exacerbations that are pauci-inflammatory vs. inflammatory at the time of enrollment.

SECONDARY OUTCOMES:
Rate of exacerbations | 1 year post hospitalization
  Number of exacerbations in the year following index admission between those with and without diastolic dysfunction.
Differences in COPD Assessment Test (CAT) in those with and without diastolic dysfunction | at or after 35 days post hospitalization
  The CAT questionnaire consists of 8 simple questions which are graded from 0 to 5. The total score can range from 0 to 40. This measure will be compared between those with and without diastolic dysfunction at the follow-up visit.
Differences in dyspnea using the modified Medical Research Council (mMRC) scale | at or after 35 days post hospitalization
  Dyspnea will be assessed using the modified Medical Research Council (mMRC) scale, ranging from 0 for minimal to 4 for severe dyspnea. We will also assess dyspnea using the more sensitive San Diego Shortness Of Breath Questionnaire (SOBQ), which rates dyspnea associated with activities of daily living (range 0 to 120). These measures will be compared between those with and without diastolic dysfunction at the follow-up visit.
Differences in dyspnea using the San Diego Shortness of Breath Questionnaire (SOBQ) | at or after 35 days post hospitalization
  Dyspnea will be assessed using the San Diego Shortness Of Breath Questionnaire (SOBQ), which rates dyspnea associated with activities of daily living (range 0 to 120). These measures will be compared between those with and without diastolic dysfunction at the follow-up visit.
Differences in 6-minute walk distance | at or after 35 days post hospitalization.
  This measure of exercise capacity will be compared between those with and without diastolic dysfunction at the follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Surya P Bhatt, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No